CLINICAL TRIAL: NCT04635319
Title: Prevalence of Facial Asymmetry Among PreOrthodontic Adult Patients: A Crosssectional Retrospective Study
Brief Title: Prevalence of Facial Asymmetry Among Orthodontic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed AbdAllah Zaki Elsayed, Mohamed Abdallah Zaki Elsayed, Cairo University
Other Study IDs: CEBD-CU-2019-05-15
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Facial Asymmetry
MeSH Terms: conditions — Facial Asymmetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18-40 years old of both sexes: patient from 18 to 40 years old seeking orthodontic treatment

SUMMARY:
To estimate the prevalence of facial asymmetry

DETAILED DESCRIPTION:
The objectives of the present study are:

* To estimate the prevalence of facial asymmetry among Egyptian population, according to type, sex, and age.
* To provide an insight into the key aspects to be taken into consideration while accomplishing an accurate diagnosis and formulation of rational integrated orthodontic-surgical treatment plan that considers correction of all aspects of the asymmetry.

ELIGIBILITY:
Inclusion Criteria:

* between 18-40 years old of both sexes who asked for orthodontic treatment

Exclusion Criteria:

* • No previous orthodontic treatment.

  * photographs of poor quality.
  * Any hereditary diseases or syndromes such as Down's syndrome or cleidocranial dysostosis.
  * Any disease of the jaw that might have affected the normal growth of permanent dentition.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Only patient's age between 18-40 years old of both sexes who asked for orthodontic treatment will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2020-11-20 (Estimated); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Type of facial asymmetry | Just before the orthodontic treatment
  chin deviation,deviation of the nasal pyramid and degree of occlusal plane cant and the relation between each type and existing malocclusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Cairo university, Cairo, Egypt